CLINICAL TRIAL: NCT00911937
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Multicenter Trial To Evaluate The Efficacy And Safety Of A Fesoterodine Flexible Dose Regimen In Patients With Symptoms Of Overactive Bladder Including Nocturnal Urinary Urgency.
Brief Title: A Trial To Evaluate The Efficacy And Safety Of Fesoterodine In Patients With Symptoms Of Overactive Bladder Including Nocturnal Urinary Urgency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0221048
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Overactive Bladder
Keywords: incontinence OAB urgency nocturia
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fesoterodine (Experimental)
  Interventions: Drug: Fesoterodine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fesoterodine — Fesoterodine 4mg and 8 mg tablets taken daily.
  Arms: Fesoterodine
Drug: Placebo — Placebo sham 4mg and 8 mg tables taken daily.
  Arms: Placebo

SUMMARY:
This study is designed to assess the efficacy of a flexible dose regimen of fesoterodine on micturition related nocturnal urgency episodes.

ELIGIBILITY:
Inclusion Criteria:

* Mean urinary frequency of >=8 micturitions per 24 hours as verified by the screening bladder diary prior to Start of Placebo run in visit (Visit 2)
* Mean number of micturition related urgency episodes >=3 per 24 hours as verified by the screening bladder diary prior to Start of Placebo run in /Visit 2 (Urgency episodes are defined as those with Urinary Sensation Scale rating >=3)
* Mean number of micturition related nocturnal urgency episodes >=2 but no more than 8 episodes per 24 hours as verified by the bladder diary at Visit 2 (nocturnal urgency episodes are defined as those with Urinary Sensation Scale rating of >3 recorded in the bed time section of the bladder diary)

Exclusion Criteria:

* A known recent history or previous diagnosis of any sleep disorder such as obstructive sleep apnea, primary insomnia, periodic limb movement, parasomnia
* Nocturia due to other underlying uncontrolled conditions, such as congestive heart failure, diabetes mellitus, diabetes insipidus, polyuria of any cause, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 963 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (102):
- United States (102):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Goodyear, Arizona
  - Pfizer Investigational Site, Litchfield Park, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Tarzana, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Dover, Delaware
  - Pfizer Investigational Site, Bonita Springs, Florida
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, DeFuniak Springs, Florida
  - Pfizer Investigational Site, Destin, Florida
  - Pfizer Investigational Site, Leesburg, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Coeur d'Alene, Idaho
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, West Des Moines, Iowa
  - Pfizer Investigational Site, Newton, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Annapolis, Maryland
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, Hyannis, Massachusetts
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, New Bedford, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Hamilton, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Kingston, New York
  - Pfizer Investigational Site, Manlius, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Burlington, North Carolina
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Concord, North Carolina
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Westerville, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Bala-Cynwyd, Pennsylvania
  - Pfizer Investigational Site, Bridgeville, Pennsylvania
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, East Greenwich, Rhode Island
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Mountlake Terrace, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Menomonee Falls, Wisconsin

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221048

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to fesoterodine 4 milligram (mg) oral tablet once daily for 4 weeks followed by placebo matched to fesoterodine 8 mg once daily depending on dose escalation as per investigator's discretion for remaining 8 weeks.
- Fesoterodine: Fesoterodine 4 mg oral tablet once daily for 4 weeks followed by dose-escalation to 8 mg once daily depending on investigator's discretion for remaining 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Fesoterodine
Started | 487 | 476
Treated | 474 | 463
Completed | 400 | 381
Not Completed | 87 | 95
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 8 | 5
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Withdrawn due to pregnancy | 1 | 0
Not completed — Adverse Event | 11 | 25
Not completed — Lack of Efficacy | 11 | 6
Not completed — Did not meet inclusion criteria | 9 | 11
Not completed — Protocol Violation | 14 | 23
Not completed — Randomized but not treated | 13 | 13
Not completed — Other | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fesoterodine | Total
Number analyzed (Participants) | 474 | 463 | 937
Age, Customized [Number; unit: participants]
  18 to 44 years | 74 | 84 | 158
  45 to 64 years | 257 | 214 | 471
  At least 65 years | 143 | 165 | 308
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 312 | 313 | 625
  Male | 162 | 150 | 312

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Micturition-related Nocturnal Urgency Episodes Per 24 Hours
Description: Micturition-related nocturnal urgency episodes had urinary sensation scale (USS) rating of 3 or more that occurred between time participant went to bed and time he or she arose to start next day. Number of nocturnal micturition-related urgency episodes per 24 hours was calculated as sum of all nocturnal micturition-related urgency episodes divided by total number of diary days collected at that visit.
Time Frame: Baseline
Population: Full analysis set (FAS): all participants who received at least 1 dose of study drug and had at least baseline or a post-baseline efficacy assessment. Here, 'N'(number of participants analyzed) signifies those participants who had baseline nocturnal urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
episodes per 24 hours | 2.93 (0.98) | 2.91 (0.90)

2. Primary Outcome: Change From Baseline in Mean Number of Micturition-related Nocturnal Urgency Episodes Per 24 Hours at Week 12
Description: Micturition-related nocturnal urgency episodes had USS rating of 3 or more that occurred between time participant went to bed and time he or she arose to start next day. Number of nocturnal micturition-related urgency episodes per 24 hours was calculated as sum of all nocturnal micturition-related urgency episodes divided by total number of diary days collected at that visit.
Time Frame: Baseline and Week 12
Population: FAS population. Last observation carried forward (LOCF) method was used to impute missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
episodes per 24 hours | -1.06 (0.06) | -1.29 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Analysis of covariance (ANCOVA) model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0030, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.22, 95% CI 2-sided [-0.37 to -0.08], Standard Error of Mean 0.08

3. Secondary Outcome: Change From Baseline in Mean Number of Micturition-related Nocturnal Urgency Episodes Per 24 Hours at Week 4
Description: Micturition-related nocturnal urgency episodes had USS rating of 3 or more that occurred between time participant went to bed and time he or she arose to start next day. Number of micturition-related nocturnal urgency episodes per 24 hours was calculated as sum of all nocturnal micturition-related urgency episodes divided by total number of diary days collected at that visit.
Time Frame: Baseline and Week 4
Population: FAS population included all participants who received at least 1 dose of study drug and had at least baseline or a post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 4.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 443 | 415
episodes per 24 hours | -0.70 (0.05) | -0.83 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0772, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.13, 95% CI 2-sided [-0.27 to 0.01], Standard Error of Mean 0.07

4. Secondary Outcome: Percent Change From Baseline in Micturition-related Nocturnal Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Percent change of micturition-related nocturnal urgency episodes per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4 and 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
percent change
  Change at Week 4 | -24.1 (38.1) | -28.4 (38.7)
  Change at Week 12 | -36.2 (37.8) | -44.5 (39.7)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 12: Ranked ANCOVA model with terms for treatment and center with ranked baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0001, Ranked ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Testing for percent change from baseline was only carried out for given endpoint if corresponding numeric change result was statistically significant

5. Secondary Outcome: Number of Nocturnal Micturitions Per 24 Hours
Description: Nocturnal micturitions were defined as micturitions with USS rating 1-5 that occurred between the time the participant went to bed and the time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The mean number of nocturnal micturitions per 24 hours was calculated as the total number of nocturnal micturitions divided by the total number of diary days collected at that visit.
Time Frame: Baseline
Population: FAS population. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal micturition frequency greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
micturitions per 24 hours | 3.19 (1.05) | 3.15 (0.99)

6. Secondary Outcome: Change From Baseline in Number of Nocturnal Micturitions Per 24 Hours at Week 4 and 12
Description: as for outcome 5
Time Frame: Baseline, Week 4 and 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal micturition frequency greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: micturitions per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
micturitions per 24 hours
  Change at Week 4 | -0.48 (0.05) | -0.59 (0.05)
  Change at Week 12 | -0.84 (0.05) | -1.02 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4: ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0827, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.12, 95% CI 2-sided [-0.25 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 12: ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0112, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least Squares mean difference = -0.19, 95% CI 2-sided [-0.33 to -0.04], Standard Error of Mean 0.07

7. Secondary Outcome: Percent Change From Baseline in Nocturnal Micturitions Per 24 Hours at Week 4 and 12
Description: Percent change of nocturnal micturitions per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
percent change
  Change at Week 4 | -15.1 (33.1) | -18.9 (31.8)
  Change at Week 12 | -26.2 (35.7) | -32.2 (35.6)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0023, Ranked ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; [statistical method as in outcome 4, analysis 1]

8. Secondary Outcome: Mean Number of Micturitions Per 24 Hours
Description: Micturitions include episodes of voluntary micturition and episodes of Urgency Urinary Incontinence [UUI]. UUI episodes were defined as those micturitions with USS rating of 5 in the diary in participants with UUI at baseline. USS rating 5: Unable to hold; leak urine.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least baseline or a post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had baseline micturition frequency greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
micturitions per 24 hours | 12.33 (3.58) | 12.30 (3.26)

9. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 4 and 12
Description: Micturitions include episodes of voluntary micturition and episodes of UUI. UUI episodes were defined as those micturitions with USS rating of 5 in the diary in participants with UUI at baseline. USS rating 5: Unable to hold; leak urine.
Time Frame: Baseline, Week 4 and 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline micturition frequency greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: micturitions per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
micturitions per 24 hours
  Change at Week 4 | -0.90 (0.11) | -1.35 (0.11)
  Change at Week 12 | -1.86 (0.13) | -2.42 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0026, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.45, 95% CI 2-sided [-0.74 to -0.16], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.0014, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.56, 95% CI 2-sided [-0.90 to -0.22], Standard Error of Mean 0.17

10. Secondary Outcome: Percent Change From Baseline in Micturitions Per 24 Hours at Week 4 and 12
Description: Percent change of micturitions per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
percent change
  Change at Week 4 | -6.7 (17.8) | -10.3 (17.7)
  Change at Week 12 | -14.2 (21.3) | -18.7 (20.0)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4: Ranked ANCOVA model with terms for treatment and center with ranked baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0016, Ranked ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0004, Ranked ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; [statistical method as in outcome 4, analysis 1]

11. Secondary Outcome: Number of Micturition-related Urgency Episodes Per 24 Hours
Description: The mean number of micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with USS rating of greater than or equal to 3 divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least baseline or a post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had baseline urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
episodes per 24 hours | 10.04 (4.01) | 9.84 (3.62)

12. Secondary Outcome: Change From Baseline in Number of Micturition-related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: as for outcome 11
Time Frame: Baseline, Week 4 and 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
episodes per 24 hours
  Change at Week 4 | -1.59 (0.16) | -2.18 (0.17)
  Change at Week 12 | -2.72 (0.18) | -3.50 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0072, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.59, 95% CI 2-sided [-1.03 to -0.16], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.0009, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.79, 95% CI 2-sided [-1.25 to -0.32], Standard Error of Mean 0.24

13. Secondary Outcome: Percent Change From Baseline in Micturition-related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Percent change of micturition-related urgency episodes per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
percent change
  Change at Week 4 | -14.9 (33.9) | -20.0 (37.2)
  Change at Week 12 | -25.7 (35.8) | -34.2 (42.3)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.0041, Ranked ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, Ranked ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; [statistical method as in outcome 4, analysis 1]

14. Secondary Outcome: Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours
Description: UUI episodes were defined as those with the USS rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least baseline or a post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had baseline UUI episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 184 | 157
episodes per 24 hours | 2.23 (2.49) | 2.20 (2.55)

15. Secondary Outcome: Change From Baseline in Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 4 and 12
Description: as for outcome 14
Time Frame: Baseline, Week 4 and 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline UUI episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 184 | 157
episodes per 24 hours
  Change at Week 4 | -0.76 (0.12) | -0.90 (0.13)
  Change at Week 12 | -1.08 (0.11) | -1.26 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.3954, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.14, 95% CI 2-sided [-0.47 to 0.19], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.2166, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.19, 95% CI 2-sided [-0.48 to 0.11], Standard Error of Mean 0.15

16. Secondary Outcome: Percent Change From Baseline in of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 4 and 12
Description: Percent change of UUI episodes per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 184 | 157
percent change
  Change at Week 4 | -34.2 (90.0) | -34.8 (102.6)
  Change at Week 12 | -58.2 (103.9) | -59.2 (71.3)

17. Secondary Outcome: Nocturnal Frequency-urgency Sum Rating Per 24 Hours
Description: Frequency-urgency sum is total USS ratings recorded for all nocturnal micturitions in 24-hour day. Number of USS ratings per 24 hours is sum of all USS ratings divided by the total diary days collected at that visit. USS scale: 1=No feeling of urgency to 5=Unable to hold: leak urine. Numerical decrease indicates improvement.
Time Frame: Baseline
Population: FAS population. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal frequency-urgency sum rating greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 441 | 420
units on a scale | 10.91 (4.14) | 10.60 (3.74)

18. Secondary Outcome: Change From Baseline in Nocturnal Frequency-urgency Sum Rating Per 24 Hours at Week 4 and 12
Description: as for outcome 17
Time Frame: Baseline, Week 4 and 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal frequency-urgency sum rating greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 441 | 420
units on a scale
  Change at Week 4 | -2.07 (0.17) | -2.46 (0.18)
  Change at Week 12 | -3.36 (0.18) | -4.08 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1018, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.39, 95% CI 2-sided [-0.85 to 0.08], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.0027, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.73, 95% CI 2-sided [-1.20 to -0.25], Standard Error of Mean 0.24

19. Secondary Outcome: Frequency-urgency Sum Rating Per 24 Hours
Description: Frequency-urgency sum is total USS ratings recorded for all micturitions in 24-hour day. Number of USS ratings per 24 hours is sum of all USS ratings divided by the total diary days collected at that visit. USS scale: 1=No feeling of urgency to 5=Unable to hold: leak urine.
Time Frame: Baseline
Population: FAS population. Here, 'N' (number of participants analyzed) signifies those participants who had baseline frequency-urgency sum rating greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
units on a scale | 39.54 (13.83) | 38.73 (12.32)

20. Secondary Outcome: Change From Baseline in Frequency-urgency Sum Rating Per 24 Hours at Week 4 and 12
Description: Frequency-urgency sum is total USS ratings recorded for all micturitions in 24-hour day. Number of USS ratings per 24 hours is sum of all USS ratings divided by the total diary days collected at that visit. USS scale: 1=No feeling of urgency to 5=Unable to hold: leak urine. Numerical decrease indicates improvement.
Time Frame: Baseline, Week 4 and 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline frequency-urgency sum rating greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 421
units on a scale
  Change at Week 4 | -4.88 (0.46) | -6.44 (0.48)
  Change at Week 12 | -8.69 (0.51) | -11.12 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0131, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -1.56, 95% CI 2-sided [-2.79 to -0.33], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.0004, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -2.43, 95% CI 2-sided [-3.78 to -1.08], Standard Error of Mean 0.69

21. Secondary Outcome: Mean Voided Volume Per Nocturnal Micturition
Description: Mean voided volume per nocturnal micturition was calculated as sum of voided volume during bedtime divided by the total number of bedtime micturition episodes with a recorded voided volume greater than 0 at that visit.
Time Frame: Baseline
Population: FAS population. Here, 'N' (number of participants analyzed) signifies those participants who had baseline voided volume per nocturnal micturition greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 369 | 345
milliliter (mL) | 172.53 (95.47) | 173.14 (95.50)

22. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Nocturnal Micturition at Week 12
Description: as for outcome 21
Time Frame: Baseline and Week 12
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 369 | 345
mL | 15.49 (5.43) | 16.81 (5.65)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8547, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = 1.32, 95% CI 2-sided [-12.82 to 15.46], Standard Error of Mean 7.20

23. Secondary Outcome: Mean Voided Volume Per Micturition
Description: Mean voided volume per micturition was calculated as sum of voided volume divided by the total number of total micturition episodes with a recorded voided volume greater than 0 at that visit.
Time Frame: Baseline
Population: FAS population. Here, 'N' (number of participants analyzed) signifies those participants who had baseline voided volume per micturition greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 396 | 372
mL | 154.56 (65.87) | 158.38 (67.40)

24. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 396 | 372
mL | 5.51 (3.17) | 4.65 (3.32)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8396, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -0.85, 95% CI 2-sided [-9.14 to 7.44], Standard Error of Mean 4.22

25. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score
Description: OAB-q: a self-administered, 33-item, questionnaire that assesses how much the participant has been bothered by selected bladder symptoms. Each item rated by participant on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Symptom bother score derived as sum of scores for questions 1-8; lowest possible raw score: 8; highest possible score: 48. Data analyzed based on transformation of the score to a 0 to 100 scale [(Actual total raw score - lowest possible value of raw score)/range]*100. Higher scores values indicative of greater symptom bother.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least baseline or a post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 416 | 395
units on a scale | 50.46 (19.54) | 48.84 (19.33)

26. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score at Week 4 and 12
Description: as for outcome 25
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 25
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 416 | 395
units on a scale
  Change at Week 4 | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4. | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4.
  Change at Week 12 | -15.91 (0.94) | -20.28 (0.97)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.0006, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = -4.37, 95% CI 2-sided [-6.84 to -1.89], Standard Error of Mean 1.26

27. Secondary Outcome: Health Related Quality of Life (HRQL) Domain and Total Score of Overactive Bladder Questionnaire (OAB-q)
Description: OAB-q: self-administered, 33-item, questionnaire, assesses how much participant has been bothered by selected bladder symptoms. Each item rated on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Questions 9 to 33 constitute HRQL, includes domains: concern, coping, sleep, and social function. HRQL domain and total raw score derived as sum of scores. Transformed score range 0 to 100 (Total HRQL or domain) = [(Highest possible raw score-Actual total raw score)/Raw score range]*100. Higher transformed scores indicative of better HRQL.
Time Frame: Baseline
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 416 | 393
units on a scale
  Concern domain | 63.29 (24.66) | 64.30 (23.08)
  Coping domain | 62.19 (26.51) | 62.26 (26.12)
  Sleep domain | 47.45 (23.25) | 49.65 (23.04)
  Social interaction domain | 82.22 (21.36) | 82.48 (20.09)
  Total | 63.56 (21.56) | 64.37 (20.61)

28. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL) Domain and Total Score of Overactive Bladder Questionnaire (OAB-q) at Week 4 and 12
Description: as for outcome 27
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 416 | 393
units on a scale
  Change at Week 4: concern domain | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4. | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4.
  Change at Week 4: coping domain | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4. | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4.
  Change at Week 4: sleep domain | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4. | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4.
  Change at Week 4: social interaction domain | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4. | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4.
  Change at Week 4: total | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4. | NA (NA) — Data was not analyzed because as per protocol OAB-q was not administered at Week 4.
  Change at Week 12: concern domain | 14.63 (1.00) | 18.05 (1.04)
  Change at Week 12: coping domain | 15.17 (1.01) | 18.32 (1.04)
  Change at Week 12: sleep domain | 18.97 (1.13) | 22.45 (1.17)
  Change at Week 12: social interaction domain | 8.27 (0.69) | 10.13 (0.72)
  Change at Week 12: total | 14.39 (0.87) | 17.42 (0.91)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 12: Concern domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0110, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = 3.42, 95% CI 2-sided [0.79 to 6.05], Standard Error of Mean 1.34
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 12: Coping domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0200, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = 3.14, 95% CI 2-sided [0.50 to 5.79], Standard Error of Mean 1.35
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Change at Week 12: Sleep domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0218, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = 3.48, 95% CI 2-sided [0.51 to 6.45], Standard Error of Mean 1.51
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Change at Week 12: Social interaction domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0458, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = 1.86, 95% CI 2-sided [0.03 to 3.68], Standard Error of Mean 0.93
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Change at Week 12: Total- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0100, ANCOVA — Statistical testing, two-sided, was done at alpha = 0.05 level; Least squares mean difference = 3.02, 95% CI 2-sided [0.72 to 5.32], Standard Error of Mean 1.17

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Fesoterodine
Serious Adverse Events (participants affected / at risk) | 9/474 | 5/463
Other Adverse Events (participants affected / at risk) | 148/474 | 187/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=474) | Fesoterodine (N=463)
Retinal detachment (Eye disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Septic arthritis staphylococcal (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=474) | Fesoterodine (N=463)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 1
Dry eye (Eye disorders) | 2 | 9
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 7 | 15
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Dry mouth (Gastrointestinal disorders) | 36 | 98
Dyspepsia (Gastrointestinal disorders) | 2 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faeces hard (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 6
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 5
Feeling abnormal (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 2
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Infected bites (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 3
Kidney infection (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 4
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 8 | 6
Tonsillitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 5
Urinary tract infection (Infections and infestations) | 8 | 9
Vaginitis bacterial (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 2
Body temperature increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Pica (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 6
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 11
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 4 | 1
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 2
Initial insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 5
Dysuria (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 3
Urine flow decreased (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.